CLINICAL TRIAL: NCT01848340
Title: An Open Label, Non-Randomized, Mass Balance Study to Investigate the Recovery, Excretion, and Pharmacokinetics of 14C-GSK1265744 Administered as a Single Oral Dose and a Placebo-Controlled, Randomized Study to Describe the Pharmacokinetics of a Supratherapeutic Dose of GSK1265744 in Healthy Adult Subjects
Brief Title: An Study to Investigate the Recovery, Excretion, and Pharmacokinetics of 14C-GSK1265744 Administered as a Single Oral Dose and a Study to Describe the Pharmacokinetics of a Supratherapeutic Dose of GSK1265744 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 117008
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-10

CONDITIONS: HIV-associated Lipodystrophy Syndrome
Keywords: mass balance; GSK1265744; supratherapeutic; integrase inhibitor; healthy volunteer
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome | interventions — cabotegravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: 14C-GSK1265744 Arm (Experimental): Each subject will receive a single 30 mg oral solution dose of GSK1265744 containing 14C-GSK1265744 of approximately 70 mcgCi (0.96 MSv) of radioactivity.
  Interventions: Drug: GSK1265744B (sodium salt) containing 14C-GSK1265744B
- Part B: GSK1265744 Arm (Experimental): In Part B - 8 subjects will be randomised to receive a single dose of GSK1265744 150 mg
  Interventions: Drug: 150 mg GSK1265744B
- Part B: Placebo Arm (Placebo Comparator): In Part B - 2 subjects will be randomised to receive a single dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1265744B (sodium salt) containing 14C-GSK1265744B — A white to slightly colored nonsterile crystalline powder for oral solution
  Arms: Part A: 14C-GSK1265744 Arm
Drug: 150 mg GSK1265744B — This is GSK1265744B (sodium salt of GSK1265744), lactose monohydrate, Microcrystalline cellulose, hypromellose, sodium lauryl sulfate, croscarmellose sodium, magnesium stearate, Opadry film-coating, white OY-S-28876 tablet
  Arms: Part B: GSK1265744 Arm
Drug: Placebo — Microcrystalline cellulose, Opadry film-coating, white OY-S-28876 tablet
  Arms: Part B: Placebo Arm

SUMMARY:
This will be a two-part study in healthy adults. Part A is a phase 1, non-randomized, open label, single-dose, single-centre mass balance study utilizing a radiolabeled dose to investigate the recovery, excretion, and pharmacokinetics of oral GSK1265744 in a cohort of 6 healthy adult male subjects. Subjects will undergo a pre-study screening visit within 30 days of the first dose and those who successfully pass pre-study assessments and meet eligibility criteria will be enrolled into the study to receive the equivalent of a 30 mg dose of GSK1265744 as an oral solution, containing approximately 70 microcuries (mcg Ci) [0.96 millisieverts (mSv)] of radioactivity under fasted conditions. Blood, urine and fecal samples will be collected for a maximum of 504 hours (21 days) following study drug administration. In Part B, approximately 10 healthy male and female subjects will be enrolled to evaluate the single-dose safety, tolerability and PK of supratherapeutic dose of GSK1265744 150 mg compared with placebo. Each subject will receive a single dose of GSK1265744 150 mg or placebo on Day 1 under fasting conditions in the morning. Blood, urine and fecal samples will be collected for 336 hours (14 days) following dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Part A: Male subjects between 30 and 55 years of age at the time of signing the informed consent.
* Part B: Male or female between 18 and 60 years of age inclusive, at the time of signing the informed consent.
* Parts A and B male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in protocol. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication.
* Part B: A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, bilateral salpingo-oophorectomy or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. Woman with child-bearing potential and is abstinent or agrees to use one of the contraception methods listed in protocol for an appropriate period of time prior to the start of dosing. Female subjects must agree to use contraception until 14 days after the last dose of study medication
* Alanine aminotransferase (ALT), alkaline phosphatase (ALP) and bilirubin <= 1.5xUpper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Body weight >= 50 kilogram (kg) and body mass index (BMI) within the range 18.5-31.0 kg/meter square (m^2) (inclusive).
* Capable of giving written informed consent
* Part A only: Available to complete the study (maximum of 21 days confinement in the clinical research unit).
* Part A only: A history of regular bowel movements (averaging one or more bowel movements per day).

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome).
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces [360 millilitre (mL)] of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor contraindicates their participation.
* Part A only: Subjects who have received a total body radiation dose of greater than 5.0 mSv or exposure to significant radiation (e.g. serial X-ray or computerised topography (CT) scans, barium meal etc.) in the 12 months prior to this study.
* Part A only: Any condition that could interfere with the accurate assessment and recovery of radioactivity [14C].
* Part A only: Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months.
* Part A only: Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy must be excluded.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Part B only: Pregnant or lactating females as determined by positive serum or urine Human Chorionic Gonadotropin (hCG) test at screening or prior to dosing.
* The subject's systolic blood pressure is outside the range of 90-140 millimetre of mercury (mmHg), or diastolic blood pressure is outside the range of 45-90 mmHg.
* History of clinically significant cardiovascular disease including: Heart rate <45 and >100 beats per minute in males and <50 and >100 beats per minute in females. QRS duration >120 milliseconds (msec) and corrected QT interval (QTc) interval B >450 msec in both males and females. Evidence of previous myocardial infarction, history/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease, any conduction abnormality [including but not specific to left or right complete bundle branch block, atrioventricular (AV) block [2nd degree (type II) or higher], Wolf Parkinson White [WPW] syndrome) or sinus pauses >3 seconds.
* Any significant arrhythmia which, in the opinion of the principal Investigator and GSK Medical Monitor, will interfere with the safety for the individual subject. Nonsustained (>=3 consecutive ventricular ectopic beats) or sustained ventricular tachycardia
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Part A: Percent recovery of total radioactive [14C] GSK1265744 in urine and feces. | Up to 21 days
  Measurement of total radioactivity present in individual samples (plasma, urine, and feces) collected for a minimum of 336 hours (14 days) post dose up to a maximum of 504 hours (21 days).
Part A: Composite of plasma GSK1265744 PK parameters to access total radioactivity in blood | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 288, 312 and 336 hours post dose.
  The PK parameters will include: Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a profile [AUC (0-t)], Area under the concentration-time curve from time zero (predose) extrapolated to infinite time [AUC (0-infinity)], Maximum observed concentration (Cmax), Time of occurrence of Cmax (tmax), Terminal phase elimination rate constant (lambda z), apparent terminal phase half-life (t1/2), and oral clearance (CL/F) of plasma GSK1265744 and total radioactivity in plasma and blood following single dose.
Part B: Number of participants with the use of concurrent medication as a measure of safety and tolerability | Up to 14 days
Part B: Absolute values and changes over time of hematology as a measure of safety and tolerability. | Up to 14 days
Part B: Absolute values and changes over time of clinical chemistry as a measure of safety and tolerability. | Up to 14 days
Part B: Absolute values and changes over time of urinalysis as a measure of safety and tolerability. | Up to 14 days
Part B: Absolute values and changes over time of vital signs as a measure of safety and tolerability. | Up to 14 days
Part B: Absolute values and changes over time of ECG intervals and ECG rhythm as a measure of safety and tolerability. | Up to 14 days
Part B: Number of participants with adverse events as a measure of safety and tolerability | Up to 14 days
Part B: Composite of plasma GSK1265744 PK parameters | Up to 14 days
  Plasma GSK1265744PK parameters following a single-dose administration of 150 mg under fasted conditions will include: AUC (0-t)], AUC (0-infinity), Cmax, tmax, lambda z, t1/2, and oral clearance (CL/F) of plasma

SECONDARY OUTCOMES:
Part A: Blood: Plasma ratio of total drug-related material (radioactivity) | Up to 21 days
  The blood: plasma ratio of total radioactivity (Cb/Cp) will be calculated at each time point by Clinical Statistics at GSK.
Part A: Percent of total radioactivity associated with red blood cells | Up to 21 days
  Percent of total radioactivity associated with red blood cells will be calculated based on radioactivity concentration in plasma and blood and hematocrit count.
Part A: Absolute values and changes over time of hematology as a measure of safety and tolerability. | Up to 21 days
Part A: Absolute values and changes over time of clinical chemistry as a measure of safety and tolerability. | Up to 21 days
Part A: Absolute values and changes over time of urinalysis as a measure of safety and tolerability. | Up to 21 days
Part A: Absolute values and changes over time of vital signs as a measure of safety and tolerability. | Up to 21 days
Part A: Absolute values and changes over time of ECG intervals and ECG rhythm as a measure of safety and tolerability. | Up to 21 days
Part A: Number of participants with adverse events as a measure of safety and tolerability | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States